CLINICAL TRIAL: NCT01398657
Title: Cryotherapy With or Without Short-term Adjuvant Androgen-Deprivation Therapy for High-Risk Localized Prostate Cancer - Open-Label Randomized Clinical Study
Brief Title: Cryotherapy With or Without Short-term Adjuvant Androgen-Deprivation Therapy in Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201103057MB
Record Dates: First submitted 2011-07-14; First posted 2011-07-20 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: localized; High risk; Prostate Cancer; Randomized; Cryotherapy; Cryoablation; Adjuvant; Androgen Deprivation Therapy; Hormone therapy; ADT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant Androgen-Deprivation Therapy (Experimental): Cryotherapy with Short-term Adjuvant Androgen-Deprivation Therapy
  Interventions: Drug: Adjuvant Androgen-Deprivation Therapy
- No adjuvant therapy (No Intervention): Cryotherapy without any adjuvant therapy

INTERVENTIONS:
Drug: Adjuvant Androgen-Deprivation Therapy — Short-term adjuvant androgen-deprivation therapy
  Other Names: Adjuvant hormone therapy
  Arms: Adjuvant Androgen-Deprivation Therapy

SUMMARY:
This is an open-label randomized clinical study comparing primary prostate cryoablation alone (No-ADT group) with cryoablation plus short-term adjuvant androgen-deprivation therapy (Adj-ADT group) in the treatment of patients with high-risk localized prostate cancer.

DETAILED DESCRIPTION:
Subjects (N=182) who have high-risk prostate cancer and have undergone primary prostate cryotherapy will be screened and randomized in a 1:1 ratio to receive either adjuvant ADT (Adj-ADT) or No-ADT until disease progression. Screening and randomization will be done within four weeks after cryoablation. Only those who are assigned to Adj-ADT will receive ADT for a total of 12 months. PSA will be checked every 3 months in the first year after Cryo and every 6 months thereafter. Long-term follow-up parameters include serum PSA and protocol-mandated biopsies (at 36 months after Cryo, irrespective of PSA levels if recurrence has not been documented). For-cause biopsy will also be done if post-Cryo PSA elevation reaches the Phoenix criteria (Nadir + 2 ng/ml) or when the treating physician thinks it necessary to document tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age>20 years
2. Histopathology proven prostate adenocarcinoma
3. Non-metastatic localized disease
4. Prostate cancer is deemed high-risk for recurrence(PSA>20 ng/ml, Gleason score>=8, or clinical staging>=T2c)
5. Subjects have undergone prostate cryoablation as the definitive treatment prior to enrolling the study
6. Subjects who have not been treated with any definitive treatments for prostate cancer, including radical prostatectomy or definitive radiotherapy. However, those who have undergone focal prostate cryoablation and have cancer recurrence are still eligible.
7. Subjects may or may not have received neoadjuvant androgen-deprivation therapy (ADT) in the forms of either castration (medical) and/or antiandrogens. Surgical castration (orchiectomy) is not allowed.
8. Subjects are willing to sign the informed consent and agree to comply with the study procedures

Exclusion Criteria:

1. Those who have been treated with > 8 weeks (collectively if not continuously) of neoadjuvant ADT prior to screening.
2. Subjects who have other cancer that is deemed not cured or are known less than 5 years except for basal cell carcinoma of the skin
3. Other conditions the investigators think may affect subject compliance or safety

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
A composite trifecta endpoint of treatment failure at 3 years after cryoablation | 3 years
  A composite trifecta endpoint of treatment failure at 3 years after cryoablation defined by either of the three, biochemical (PSA) recurrence (by the Phoenix criteria) or biopsy-proven recurrence or initiation of hormone therapy for disease recurrence whichever comes first.

SECONDARY OUTCOMES:
Time to the composite endpoint of treatment failure since cryoablation | 3 years
  Time to the composite endpoint of treatment failure since cryoablation
Biochemical (PSA) recurrence rate at 3 years | 3 years
  Biochemical (PSA) recurrence rate at 3 years
Biochemical (PSA) recurrence-free survival | 3 years
  Biochemical (PSA) recurrence-free survival
Biopsy-proven recurrence rate at 3 years | 3 years
  Biopsy-proven recurrence rate at 3 years
Biopsy-proven recurrence-free survival | 3 years
  Biopsy-proven recurrence-free survival
Safety profile | 3 years
  Hormone therapy related toxicities such as liver function alteration, libido changes, alterations in quality of life as measured by QLQ C30 and PR25 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan